CLINICAL TRIAL: NCT01067235
Title: Prospective, Randomized, Double-blind Study, Parallel-group, Multi-center Trial Assessing the Effects of Escalating Doses of BF2.649 and BF2.649 Add on Modafinil on Cataplexy in Patients With Narcolepsy
Brief Title: Efficacy and Safety Study of BF2.649 and BF2.649 Add on Modafinil on Cataplexy in Patients With Narcolespy
Acronym: Harmony2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P07-07 / BF2.649; 2008-007845-29 (EudraCT Number)
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2012-06

CONDITIONS: Narcolepsy; Cataplexy; Excessive Daytime Sleepiness
Keywords: Narcolespy; Cataplexy; Excesssive daytime Sleepiness; Sleep Disorders; Sleep attacks; Orphan Drug; Pitolisant
MeSH Terms: conditions — Narcolepsy; Cataplexy; Disorders of Excessive Somnolence; Sleep Wake Disorders | interventions — pitolisant; Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BF2.649 + Modafinil placebo (Experimental)
  Interventions: Drug: BF2.649
- BF2.649 + Modafinil (Experimental)
  Interventions: Drug: BF2.649 add on Modafinil

INTERVENTIONS:
Drug: BF2.649 — BF2.649 oral capsules at 10, 20 or 40 mg/day associated with Modafinil Placebo capsules for 8 weeks
  Other Names: Pitolisant
  Arms: BF2.649 + Modafinil placebo
Drug: BF2.649 add on Modafinil — BF2.649 oral capsules at 10, 20 or 40 mg/day associated with Modafinil capsules at 200 mg per day for 8 weeks
  Other Names: Pitolisant; Modiodal
  Arms: BF2.649 + Modafinil

SUMMARY:
The objective of this study is to evaluate and compare the efficacy and safety of escalating doses of BF2.649 and BF2.649 add on Modafinil on cataplexy in patients with narcolepsy

DETAILED DESCRIPTION:
BF 2.649, a new molecule, reduces significantly the diurnal sleepiness and demonstrated its anti-cataplexy effect in pre-clinical and clinical studies.

The objective of this POC study are firstly to evaluate and compare the efficacy and safety of escalating doses of BF2.649 and BF2.649 add on Modafinil (200 mg/day) on cataplexy attacks, and secondly to evaluate the additive/synergistic effect and safety of the combination of BF2.649 and Modafinil on EDS as assessed by both of objective and subjective measures including ESS, MWT, patients sleep diary.

ELIGIBILITY:
Inclusion Criteria:

* "De novo" patients with newly diagnosed narcolespy and cataplexy , and not taking any treatment for Excessive Daytime Sleepiness(EDS) and cataplexy
* patients with previously diagnosed narcolepsy and cataplexy and not taking any treatment for EDS and cataplexy for more than 3 months
* partial or total cataplexy attacks with a frequency of at least 5 per week during a 14 day baseline period and ESS >or= 14 at the end of the baseline period

Exclusion Criteria:

* Patients who are unable or unwilling to temporarily discontinue any no-authorized drugs or substances
* Current or recent history of a substance abuse or dependence disorder including alcohol abuse
* Psychiatric and neurological disorders such as psychosis or dementia, bipolar illness, severe anxiety, clinical depression, history of seizure disorder or other problem that in the investigator's opinion would preclude the patient's participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Cataplexy attacks reported on sleep diary | every days from screening visit (day-14) to final visit (day 56)

SECONDARY OUTCOMES:
Sleep Diary: number and duration of diurnal sleep and sleepiness episodes, | every days from screening visit (day-14) to final visit (day 56)
Maintenance of Wakefulness Test (MWT), Test of Sustained Attention to Response Task (SART). | at inclusion and after 8-week treatment
Epworth Sleepiness Scale (ESS) | at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Bassetti, Principal Investigator — Neurocenter of Southern Switzerland,Lugano
Locations (1):
- Neurocenter (EOC) of Southern Switzerland, Lugano, Switzerland